CLINICAL TRIAL: NCT06648668
Title: A Randomized, Participant- and Investigator-blinded, Placebo-controlled, Parallel-group Study to Assess the Safety, Tolerability, and Pharmacokinetics of Oral TMP-301 Given Concurrently With Cocaine
Brief Title: A Study to Investigate the Interaction Between TMP-301 and Cocaine.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tempero Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMP-301-CUD-102
Record Dates: First submitted 2024-10-10; First posted 2024-10-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Cocaine Use Disorder
Keywords: CUD, Substance Use Disorder, SUD
MeSH Terms: conditions — Systemic carnitine deficiency; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, Participant- and Investigator-blinded, Placebo-controlled, Parallel-group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TMP-301 (Experimental): Once daily [QD] × 14 days
  Interventions: Drug: TMP-301
- Placebo (Placebo Comparator): Once daily [QD] × 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TMP-301 — Once daily [QD] × 14 days
  Arms: TMP-301
Drug: Placebo — Once daily [QD] × 14 days
  Arms: Placebo

SUMMARY:
This will be a randomized, double-blind, placebo-controlled, parallel-group study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of oral TMP-301, given concurrently with cocaine. The study will consist of 4 phases: Screening, Baseline, Treatment, and Follow-up.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled, parallel-group study to assess the safety, tolerability, PK, and PD of oral TMP-301, given concurrently with cocaine. The study will consist of 4 phases: Screening, Baseline, Treatment, and Follow-up. The Screening Phase will be completed as an outpatient visit within 24 days of the Baseline Phase and will consist of a standard medical screen. Within 24 days of a standard medical screening, eligible participants will return to the clinical site as inpatients to complete the Baseline Phase. All participants will remain in-clinic for the duration of the 7-day Treatment Phase. Following confirmation of eligibility, participants will be randomized to one of two treatment groups, either TMP-301 or. A safety follow-up visit will be conducted on Day 23.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 55 years of age, inclusive.
2. Understand the study procedures, follow instructions, and provide written informed consent.
3. Have a body mass index (BMI) within a range of 18.0 to 34.0 kg/m2 and body weight ≥50.0 kg at Screening.
4. Healthy, as determined by no clinically significant medical history, physical examination, 12-lead ECG, vital signs, and clinical laboratory results (including hematology, clinical chemistry, urinalysis, and serology) at Screening, as judged by the investigator.
5. ≥6 uses of cocaine by the smoked or IV route in the 12 months prior to Screening
6. Provide a positive urine drug screen (UDS) for cocaine at least once during the screening period or at admission. Repeat or rescheduled testing will be allowed at the investigator's discretion.
7. Have BP and Heart Rate (HR) within the following ranges after 5 minutes' rest at Screening and admission:

   1. SBP: 90 to 139 mmHg, inclusive
   2. DBP: 50 to 89 mmHg, inclusive
   3. HR: 45 to 99 bpm, inclusive
8. If male, agree to use a double-barrier method (e.g., condom and spermicide) or agree to remain abstinent from heterosexual intercourse at the time of Screening, during the study, and for 90 days following the last administration of study drug. Male participants must agree not to donate sperm during the study and for 90 days following the last administration of study drug.
9. If female, meets one of the following criteria:

   a. Physiological postmenopausal status, defined as the following: i. Absence of menses for at least 12 months prior to the first study drug administration (without an alternative medical condition); OR b. Surgically sterile (e.g., have undergone hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or tubal ligation/occlusion).

Exclusion Criteria:

1. Meet current Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition (DSM-5) criteria for any SUDs other than cocaine, cannabis, or nicotine. Diagnosis of mild to moderate alcohol use disorder will not be considered exclusionary.
2. Have a DSM-5 psychiatric disorder other than SUD, including but not limited to, Bipolar Disorder, Major Depressive Disorder, or Schizophrenia, or have a neurological disorder requiring ongoing treatment and/or making study participation unsafe.
3. Have any previous medically adverse reaction to cocaine, including loss of consciousness, chest pain, paranoid reaction, or epileptic seizure.
4. Have a 12-lead ECG with repeated demonstration of corrected QT interval (QTcF) ≥470 msec in female participants or ≥450 msec in male participants at Screening.
5. Unable to tolerate a 20 mg cocaine IV infusion (Day -2) or a 40 mg cocaine IV infusion (Day -1) during the Baseline Phase, as judged by the investigator or designee and per criteria in protocol;
6. History or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, gastrointestinal, neurological, respiratory, or endocrine disorder, which would preclude safe or successful completion of the study, as determined by an investigator.
7. Have a history of any illness, or a family history of early significant cardiovascular disease that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drugs to the participant.
8. Have a significant risk of developing psychosis (assessed by Prevention through Risk Identification, Management, and Education [PRIME] screen) or have a personal history of psychotic symptoms (hallucinations or delusions), with or without a formal psychiatric diagnosis.
9. Have a family history of significant mental, behavioral, or neurodevelopmental disorders, unless determined by the investigator to be not clinically significant (NCS).
10. Have a current or past history of seizures, including alcohol- or stimulant-related seizures (excluding childhood febrile seizures), or significant family history of idiopathic seizure disorder or clinically significant (CS) head injury.
11. Have a diagnosis of adult (i.e., 21 years or older) asthma, or chronic obstructive pulmonary disease (COPD), including those with a history of acute asthma within the past two years, and those with current or recent (past 2 years) treatment with inhaled or oral beta-agonist.
12. Smoked >40 cigarettes per day on average, in the month prior to Screening, or are unable to abstain from smoking (or use of any nicotine-containing substance) for at least 8 hours.
13. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by an investigator.
14. History of stomach or intestinal surgery, or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).
15. Evidence of CS hepatic or renal impairment, including alanine aminotransferase (ALT), aspartate aminotransferase (AST), or creatinine >1.5 × the upper limit of normal (ULN) at Screening or admission to the Baseline Phase. Retesting may be permitted at the discretion of an investigator.
16. Any clinically significant abnormalities in laboratory test results at Screening that would, in the opinion of an investigator, increase the participant's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data. Retesting may be permitted at the discretion of an investigator.
17. Are seropositive for hepatitis B surface antigen, hepatitis C antibody (asymptomatic hepatitis C virus infection at Screening is allowed), or human immunodeficiency virus (HIV).
18. Have significant current suicidal ideation or a history of suicide attempt within the past 12 months, as assessed by the C-SSRS (baseline version), or have significant current homicidal ideation.
19. If female, is currently pregnant (positive pregnancy test) or lactating, or who is planning to become pregnant within 30 days of last study drug administration.
20. Use of a prohibited medication or investigational drug, as specified in protocol.
21. Consumption of any foods or beverages that alter CYP1A2 activity (e.g., barbecued food or cruciferous vegetables, such as broccoli and cauliflower) or CYP3A4 activity (e.g., foods or beverages containing grapefruit or Seville-type oranges), within 7 days prior to admission to the Baseline Phase (a list of prohibited foods will be provided to participants).
22. Have received blood products within 2 months of admission to the Baseline Phase.
23. Positive UDS at admission to the Baseline Phase (Day -3), other than cocaine or tetrahydrocannabinol (THC). If THC is positive, a cannabis intoxication evaluation will be done by an investigator, and participants may be permitted to continue in the study at the discretion of an investigator. The UDS may be repeated and/or the participant may be rescheduled at the investigator's discretion.
24. Have donated or lost more than 500 mL whole blood within 56 days or have donated plasma within 7 days prior to Screening, or have participated in another clinical trial within the last 30 days prior to screening.
25. Have difficulty with venous access or are unsuitable or unwilling to undergo catheter insertion or direct venipuncture.
26. Currently on probation or have any pending legal action that could prohibit participation or compliance in the study.
27. Are an employee of the sponsor, a research site staff member directly affiliated with this study, or are an immediate family member, defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
28. Have any other condition that, in an investigator's opinion, (i) puts participant at increased risk, (ii) could confound the study results, (iii) may interfere significantly with participant's participation in the study, or (iv) have the potential to limit the participant's ability to complete the study .

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-01-04 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of TMP-301 alone via incidence and severity of treatment-emergent adverse events (TEAEs) with cocaine infusions. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 in combination with cocaine via incidence and severity of treatment-emergent adverse events (TEAEs) with cocaine infusions. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 alone via peak change from baseline of heart rate (CFBmax). | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 in combination with cocaine via peak change from baseline of heart rate (CFBmax). | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 alone via peak change from baseline of systolic blood pressure (SBP). | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 in combination with cocaine via peak change from baseline of systolic blood pressure (SBP). | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 alone via peak change from baseline of diastolic blood pressure (DBP). | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 in combination with cocaine via peak change from baseline of diastolic blood pressure (DBP). | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 alone via peak change from baseline of quantitative electrocardiogram PR interval | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 alone via peak change from baseline of quantitative electrocardiogram QRS complex. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 in combination with cocaine via peak change from baseline of quantitative electrocardiogram PR interval. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 in combination with cocaine via peak change from baseline of quantitative electrocardiogram QRS complex. | Baseline to Day 23

SECONDARY OUTCOMES:
To assess the maximum observed plasma concentration (Cmax) of cocaine alone. | Days 7 and 14
To assess the maximum observed plasma concentration (Cmax) of cocaine with TMP-301. | Days 7 and 14
To assess the Tmax of cocaine alone. | Days 7 and 14
To assess the Tmax of cocaine with TMP-301. | Days 7 and 14
To assess the area under the plasma concentration-time curve from time 0 to the last measured concentration (AUC0-t) of cocaine alone. | Days 7 and 14
To assess the area under the plasma concentration-time curve from time 0 to the last measured concentration (AUC0-t) of cocaine with TMP-301. | Days 7 and 14
To assess the AUC from time 0 to infinity (AUC0-inf) of cocaine alone. | Days 7 and 14
To assess the AUC from time 0 to infinity (AUC0-inf) of cocaine alone in combination with TMP-301. | Days 7 and 14
To assess the elimination rate constant (λz) of cocaine alone. | Days 7 and 14
To assess the elimination rate constant (λz) of cocaine in combination with TMP-301. | Days 7 and 14
To assess the t1/2 of cocaine alone. | Days 7 and 14
To assess the t1/2 of cocaine in combination with TMP-301. | Days 7 and 14
To assess the apparent clearance (CL; if data permit) of cocaine alone. | Days 7 and 14
To assess the apparent clearance (CL; if data permit) of cocaine in combination with TMP-301. | Days 7 and 14
To assess the apparent volume of distribution (Vd; if data permit) of cocaine alone. | Days 7 and 14
To assess the apparent volume of distribution (Vd; if data permit) of cocaine in combination with TMP-301. | Days 7 and 14
To assess the metabolite-to-parent ratio (Cmax) of cocaine alone. | Days 7 and 14
To assess the metabolite-to-parent ratio (area under the plasma concentration versus time curve) of cocaine alone. | Days 7 and 14
To assess the metabolite-to-parent ratio (Cmax) of cocaine in combination with TMP-301. | Days 7 and 14
To assess the metabolite-to-parent ratio (area under the plasma concentration versus time curve) of cocaine in combination with TMP-301. | Days 7 and 14
To assess the visual analog scale (0-100): maximum effect (Emax) from time 0 to 60 minutes post-cocaine infusion of cocaine alone. | Days 7 and 14
  Higher score is worse
To assess the visual analog scale (0-100): Area Under the Effect Curve (AUE) from time 0 to 60 minutes post-cocaine infusion of cocaine alone. | Days 7 and 14
  Higher score is worse
To assess the visual analog scale (0-100): maximum effect (Emax) from time 0 to 60 minutes post-cocaine infusion of cocaine in combination with TMP-301. | Days 7 and 14
  Higher score is worse
To assess the visual analog scale (0-100): AUE from time 0 to 60 minutes post-cocaine infusion of cocaine in combination with TMP-301. | Days 7 and 14
  Higher score is worse
To assess the Brief Substance Craving Scale (BSCS) scores over time of cocaine alone. | Days 7 and 14
  The BSCS is a self-administered assessment that asks the participant to rate his or her craving for cocaine. The BSCS used for this study is a modification of the State of Feelings and Cravings Questionnaire.
To assess the Brief Substance Craving Scale (BSCS) scores over time of cocaine in combination with TMP-301. | Days 7 and 14
  The BSCS is a self-administered assessment that asks the participant to rate his or her craving for cocaine. The BSCS used for this study is a modification of the State of Feelings and Cravings Questionnaire.
To assess the Cmax of TMP-301. | Days 7 and 14
To assess the Tmax of TMP-301. | Days 7 and 14
To assess the AUC during a dosing interval (AUC0-τ) of TMP-301. | Days 7 and 14
To assess the λz of TMP-301. | Days 7 and 14
To assess the t1/2 of TMP-301. | Days 7 and 14
To assess the CL/F (if data permit) of TMP-301. | Days 7 and 14
To assess the Vd/F (if data permit) of TMP-301. | Days 7 and 14
To evaluate the safety and tolerability of TMP-301 as assessed by the incidence and severity of Treatments Emergent Adverse Events (TEAEs). | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 as assessed by number of participants taking concomitant medications taken during study participation. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 as assessed by systolic blood pressure. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 as assessed by diastolic blood pressure. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 as assessed by heart rate. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 as assessed by electrocardiogram PR interval. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 as assessed by electrocardiogram QRS complex. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 as assessed by number of participants with abnormal laboratory test results. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 as assessed by Beck Depression Inventory (BDI) scores (0-63) over time. | Baseline to Day 23
  Score of 63 is worse.
To evaluate the safety and tolerability of TMP-301 as assessed by the Brief Psychiatric Rating Scale (BPRS) scores (0-126) over time. | Baseline to Day 23
  Score of 126 is worse.
To evaluate the safety and tolerability of TMP-301 as assessed by number of participants with abnormal physical examination findings. | Baseline to Day 23
To evaluate the safety and tolerability of TMP-301 as assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) score (0-5) | Baseline to Day 23
  Score of 5 is worse.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No